CLINICAL TRIAL: NCT06400667
Title: Development of New Multifactorial Functional Assessment Protocols and Related Indices for Pediatric Age -Functional Assessment Protocol for the Upper Limb
Brief Title: Functional Assessment Protocol for the Upper Limb for Pediatric Age
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1054
Record Dates: First submitted 2024-03-19; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Upper Extremity; Child; Range of Motion, Articular
Keywords: Kinematics; Upper limb; Motion analysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Experimental): Subjects without upper limb disease
  Interventions: Device: Upper limb Kinematic Assessment with Optoelectronic system
- Pathological subjects (Experimental): Subjects with a brain injury like cerebral phalsy or acquired brain injury
  Interventions: Device: Upper limb Kinematic Assessment with Optoelectronic system

INTERVENTIONS:
Device: Upper limb Kinematic Assessment with Optoelectronic system — All measurements will be obtained using an optoelectronic multicamera system for human motion analysis (with eight high-resolution cameras with infrared light and a sampling frequency of 60 Hz. The experimental protocol require the positioning of markers (plastic spheres covered by reflecting film, 10 mm in diameter). Markers will be placed by clinical operators (physiotherapists with training in optoelectronic system for human motion analysis) after training and experience in recognition of the position of body landmarks. During the data acquisition protocol, the subject perform five trial for each upper limb of a determinate functional task for each session. Every subject repeat this operations 2 times with 2 different operators.

SUMMARY:
During data acquisition a trained therapist placed reflective markers on the skin of the participants in the selected body landmarks. The participants will be asked to perform five trial for each upper limb of a determinate functional task for each session.

DETAILED DESCRIPTION:
Acquired brain injuries (ABIs)and cerebral palsy (CP) can lead to a wide range of impairments, including weakness or paralysis on one side of the body known as hemiplegia. In hemiplegic patients, the rehabilitation of the upper limb skills is crucial, because the recovery has an immediate impact on patient quality of life. Therefore, an accurate upper limb motion analysis may be useful during medical diagnostic-therapeutic process, it is relevant to understand the integrated and synergic motion of the upper limbs for a variety of applications, such as clinical diagnosis, endoprosthesis design, and the evaluation of treatment outcomes. There are many clinical scales used to assess the upper extremity. Most of these use an ordinal-level scoring system, with scores assigned to the patient by the observing physician or therapist. Another way to assess upper limb activity is through kinematics data from 3D motion capture. Kinematics data provide an objective and quantifiable method, as well as allowing the use of several otherwise undetectable metrics: time, velocity, and joint angles. The aim of this study is introducing a new protocol consisting of a marker set, i.e. an innovative and integrated biomechanical model of the human body for the global analysis of upper limb during functional tasks allows for a more detailed evaluation of the motor behavior and its abnormalities to better characterize the functionality of the upper, both on the sagittal, frontal and transversal plane. The development of a new protocol of analysis requires the validation before its definitive and clinical application. More in detail, the validation should be carried out in terms of both comparisons with reference absolute measures and the evaluation of its repeatability with healthy subjects.

ELIGIBILITY:
For healthy group:

Inclusion Criteria:

- absence of functional impairments in the upper limbs

Exclusion Criteria:

* behavioral, visual or auditory problems
* presence of pain in the upper limbs

For pathological group:

Inclusion Criteria:

* Unilateral PCI candidates for CIMT (Constraint Induced Movement Therapy) treatment;
* Acquired brain injury candidates for CIMT or Bimanual treatment;
* Ability to understand and follow test instructions.

Exclusion Criteria:

* behavioral, visual or auditory problems
* presence of pain in the upper limbs

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
Intra/Inter Operator Reliability | Through study completion, an average of 3 year
  In the intra and interoperator repeatability analysis the investigators considered the correlation coefficient for the average RoM (in the 5 trials) in corresponding sessions. In particular, the investigators referred to standard interpretation criteria: the ICC values 0.5 and 0.75 indicate moderate reliability, values between 0.75 and 0.9 indicate good reliability, and values greater than, 0.90 indicate excellent reliability
Measures accuracy analysis | Year 1
  For the accuracy analysis, the comparison between the reference measures and the measure obtained with the optoelectronic system for every segment of the spine was assessed through the root mean square error.
Usability assessment | Through study completion, an average of 3 year
  About the usability assessment, the System Usability Scale (SUS) collected at the end of each acquisition and calculated the average score value. The SUS provides a reliable tool for measuring the usability. The SUS questionnaire consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Andreoni, Principal Investigator — IRCCS E. Medea - La Nostra Famiglia
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy